CLINICAL TRIAL: NCT02237677
Title: Cannabinoid-1 (CB1) Receptor Positron Emission Tomography (PET) Imaging Reveals Gender Differences in Posttraumatic Stress Disorder (PTSD)
Brief Title: CB1 Receptor PET Imaging Reveals Gender Differences in PTSD
Status: Terminated | Type: Observational
Why Stopped: The original PI, Alexander Neumeister, left NYULMC. No data was analyzed.
Sponsor: NYU Langone Health (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 12-02787
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
Keywords: Post-traumatic stress disorder (PTSD); Trauma; Neuroimaging; Positron emission tomography (PET); [11C]OMAR; Endocannabinoid
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Post-traumatic stress disorder (PTSD): Post-traumatic stress disorder (PTSD)
  Interventions: Other: Positron emission tomography (PET) imaging
- Healthy Controls (HC): Healthy Controls (HC)
  Interventions: Other: Positron emission tomography (PET) imaging

INTERVENTIONS:
Other: Positron emission tomography (PET) imaging — Positron emission tomography (PET) imaging

SUMMARY:
The objective of the proposed translational study is to test a model, based upon basic science studies, exploring multisystem impairments in PTSD including endocannabinoid (eCB) and glucocorticoids in the modulation of fear memories by examining the cannabinoid type 1 (CB1) receptor in a PTSD fear circuit as well as glucocorticoid function. The investigators propose that impaired eCB signaling in PTSD resulting in the maladaptive neurobehavioral response to the stressor is associated with an upregulation of the CB1 receptors and insufficient glucocorticoid signaling.

DETAILED DESCRIPTION:
The eCB - anandamide and 2-arachidonoylglycerol (2-AG) - and their attending cannabinoid (CB) receptors which are found in high densities in a fear circuitry involving the amygdala, hippocampus, the anterior cingulate cortex and prefrontal cortex serve important functions in the regulation of stress-coping behaviors. Besides eCB regulation there is strong evidence from ongoing research of the investigators group and others suggesting an important role for glucocorticoid signaling as an endpoint of the biochemical sequelae initiated by stressful or aversive stimuli. One of the long-term research goals of our lab is to understand such functions and determine their relevance to the pathogenesis of PTSD and to provide a more integrative view on neurobiological mechanisms that are involved in the regulation of the neuroadaptive response to stress. The objective of the proposed translational study is to test a model, based upon basic science studies, exploring multisystem impairments in PTSD including eCB and glucocorticoids in the modulation of fear memories by examining the CB1 receptor in a PTSD fear circuit as well as glucocorticoid function. The investigators propose that impaired eCB signaling in PTSD resulting in the maladaptive neurobehavioral response to the stressor is associated with an upregulation of the CB1 receptors and insufficient glucocorticoid signaling.

ELIGIBILITY:
Inclusion Criteria for Patients with PTSD:

1. age 18-55 years old
2. currently diagnosed with PTSD and symptomatic with a Clinician-Administered PTSD Scale (CAPS) score > 50.

Inclusion Criteria for healthy subjects:

1. age 18-55 years old
2. no personal or first-degree family history of any Axis I diagnosis.

Exclusion criteria for Patients with PTSD:

1. any primary Axis I disorder other than PTSD (e.g. psychosis);
2. medical or neurological illnesses likely to affect physiology or anatomy, i.e. uncontrolled hypertension, cardiovascular disorders;
3. a history of drug (including benzodiazepines (BZD)) dependence (DSM IV criteria) within 1 year of the study and lasting longer than 2 years, except for alcohol dependence
4. current pregnancy (as documented by pregnancy testing at screening or on the day of PET imaging study)
5. current breast feeding
6. nicotine dependence
7. suicidal ideation or behavior
8. general MRI exclusion criteria, i.e. pacemakers, metals in the body
9. Human immunodeficiency virus (HIV) (due to possible neuropsychiatric effects);
10. use of opioid medications within 2 weeks of the PET study
11. having an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participation in the study
12. seriously claustrophobic
13. blood donation within 8 weeks prior to the study.

Exclusion criteria for healthy subjects:

1. any history or current primary Axis I disorder
2. medical or neurological illnesses likely to affect physiology or anatomy, i.e. uncontrolled hypertension, cardiovascular disorders
3. a history of drug (including benzodiazepines [BZD]) dependence (DSM IV criteria) within 1 year of the study and lasting longer than 2 years, except for alcohol dependence
4. current pregnancy (as documented by pregnancy testing at screening or on the day of PET imaging study)
5. current breast feeding
6. nicotine dependence
7. suicidal ideation or behavior
8. general MRI exclusion criteria, i.e. pacemakers, metals in the body
9. HIV (due to possible neuropsychiatric effects)
10. use of opioid medications within 2 weeks of the PET study
11. having an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participation in the study
12. seriously claustrophobic
13. blood donation within 8 weeks prior to the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects are between the age range of 18 to 55, are medically healthy and currently not taking any medications to treat any medical illness, history of post-traumatic stress disorder (PTSD) or healthy control.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Volume of distribution (VT) of cerebral CB1 receptor expression in PTSD and controls within a fear circuit of brain regions that regulate stress-related behaviors using the CB1 radioligand carbon - 11 (11C) [11C]OMAR and PET. | Two months
  To examine group differences in cerebral CB1 receptor expression in PTSD and controls within a fear circuit of cortical and subcortical brain regions that regulate stress-related behaviors using the CB1 radioligand [11C]OMAR and PET.
  Hypothesis: PTSD patients will show greater [11C]OMAR VT (i.e. CB1 binding) values than both control groups, trauma-exposed and non-trauma exposed control subjects who will not be different.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Marmar, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States